CLINICAL TRIAL: NCT01545102
Title: Assessment of Exercise Intensity in Cardiac Rehabilitation Programmes for Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy Lloyd (Other)
Responsible Party: Sponsor-Investigator, Guy Lloyd, Consultant Cardiologist, Eastbourne General Hospital
Organization: Eastbourne General Hospital (Other)
Other Study IDs: TN11-26
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac rehabilitation is the ideal comprehensive intervention for patients with chronic heart failure (CHF), since it addresses the complex interplay of medical, psychological and behavioural factors facing these individuals. Structured exercise training within a cardiac rehabilitation programme is firmly recommended for these patients. However, it is questionable whether patients are achieving an adequate dose of exercise to provide optimal benefits. The essential components for setting optimal training include the appropriate mode, duration, frequency and intensity of exercise. UK surveys of cardiac rehabilitation describe the frequency and duration of training, but here is scant information on exercise intensity. However, it is apparent that randomised controlled trials of exercise training use doses more than 4 times greater than in UK current practice. The Eastbourne Exercise Cardiology Research Group has demonstrated that although patients benefit from improved quality of life and submaximal fitness after a hospital outpatient cardiac rehabilitation programme, they do not achieve the increases in important prognostic indicators reported by the majority of exercise training trials.

The critical factor in terms of eliciting a sufficient training effect while minimising risk is the intensity of the exercise performed. It is now widely accepted that the traditional methods of using fixed percentages of maximal heart rate or oxygen uptake to set exercise intensity include serious errors. The European Society of Cardiology recommends that cardiopulmonary exercise testing should be used to provide an objective evaluation of the metabolic demand of exercise. This allows physiologically meaningful reference points to be established for aerobic exercise prescription and is the solution to defining safe and effective training intensities. The next step is to determine whether this information can be transferred to a practical cardiac rehabilitation environment to set and monitor exercise intensity

DETAILED DESCRIPTION:
Background Heart failure is a chronic, costly and life-threatening disorder that constitutes a significant burden for individuals and the National Health Service [There are 27,000 new cases reported per annum in the UK. Cardiac rehabilitation (CR) is recommended as the ideal comprehensive intervention since it addresses the complex interplay of medical, psychological and behavioural factors facing CHF patients and carers.

Study Aim Primary objective to describe the exercise intensity, defined by oxygen uptake (VO2) in terms of the individual physiological thresholds, in CHF patients undergoing CR according to current guidelines Primary end point: VO2 Secondary objectives Secondary objectives of this study are:-

1. To measure resting and exercising energy expenditure in order to a) establish the value of 1 MET (resting metabolic rate) for patients with CHF, and b) to establish the MET value (defined as multiples of resting metabolic rate) for exercises performed in CR sessions
2. To measure affective responses (feeling very bad - feeling very good; levels of energy - tiredness and tension - calmness) to exercise during CR sessions
3. To measure weekly physical activity level in CHF patients undergoing Phase III and IV CR.

For the secondary analysis the following secondary end points and parameters will be established

1. MET values, defined as multiples of resting oxygen uptake or resting metabolic rate (1 MET), for different CR exercises
2. Ratings of affective response on the Feelings Scale (FS) and ratings of perceived activation on the Felt Arousal Scale (FAS).
3. Average daily activity over 7 day period in terms of steps per day and periods spent sitting, standing and walking

ELIGIBILITY:
Inclusion criteria:

* Systolic heart failure with resting left ventricular ejection fraction below 40%
* New York Heart Association (NYHA) class I-III
* clinically stable for at least 4 weeks on optimised medication dosage according to current guidelines

Exclusion criteria:

* Acute coronary syndrome within past 6 months
* Untreated lifethreatening cardiac arrhythmias
* Acute heart failure (during initial period of haemodynamic instability)
* Uncontrolled hypertension
* Advanced atrioventricular block
* Acute myocarditis or pericarditis
* Symptomatic aortic stenosis
* Severe hypertrophic obstructive cardiomyopathy
* Acute systemic illness Intracardiac thrombus
* Progressive worsening of exercise tolerance of dyspnoea at rest over previous 35 days
* Significant ischaemia during low intensity exercise (< 2 METS, < 50W)
* Uncontrolled diabetes
* Recent embolism
* Thrombophlebitis
* New onset atrial fibrillation/flutter
* > 1.8 kg increase in body mass over previous 13 days
* Concurrent, continuous or intermittent dobutamine therapy
* Decrease in systolic blood pressure with exercise
* NYHA Functional Class IV
* Complex ventricular arrhythmia at rest or appearing with exertion
* Supine resting heart rate > 100 beats/min
* Patient is participating in a conflicting study, is unable to perform exercise testing
* Patient lacks the capacity to consent or cannot comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 21 CHF patients from Heart Failure clinic at Eastbourne District General Hospital
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the oxygen uptake(VO2)during exercise | 13 weeks

SECONDARY OUTCOMES:
Affective responses (e.g. feelings of pleasure/displeasure) | 13 weeks
  Questionnaire used to measure affective responses (Feelings Scale, Felt Anxiety Scale and Activation/Deactivation )
Weekly physical activity | 13 weeks
  Average daily physical activity: Participants' freeliving activity will be classified by ActivPAL into periods spent sitting, standing and walking, and daily energy expenditure will also be estimated from this information.

CONTACTS AND LOCATIONS:
Overall Officials: Guy W Lloyd, MD, Principal Investigator — Eastbourne General Hospital
Locations (1):
- Eastbourne General Hospital, Eastbourne, East Sussex, United Kingdom